CLINICAL TRIAL: NCT07231458
Title: A Phase I/Ib Open-Label Study of ABX-001 Administered With and Without the Anti-PD-1 Immune Checkpoint Inhibitor Pembrolizumab in Participants With Advanced Solid Tumors Who Are Beyond Standard of Care
Brief Title: A Study to Test a New Immunotherapy, ABX-001, Alone and in Combination With the Marketed Drug, Pembrolizumab, for the Treatment of Tumors Previously Treated With Other Therapies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abalos Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABX-001-01; 2024-512403-39-01 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Immunotherapy; Non-oncolytic virus; Arenavirus
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): ABX-001 is administered intravenously (IV) alone
  Interventions: Drug: ABX-001
- Part B (Experimental): ABX-001 is co-administered intravenously (IV) with pembrolizumab
  Interventions: Drug: ABX-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ABX-001 — ABX-001 administered intravenously (IV)
Drug: Pembrolizumab — Pembrolizumab administered intravenously (IV)
  Arms: Part B

SUMMARY:
This is a Phase I/Ib first-in-human, open-label, non-randomized, multicenter, multi-country study to evaluate the safety and tolerability and to establish a recommended Phase 2 dose (RP2D) as well as assess preliminary clinical activity of ABX-001 administered intravenously (IV) alone (Part A) or co-administered with pembrolizumab (Part B) in participants with refractory/relapsed advanced solid tumors.

DETAILED DESCRIPTION:
The study will consist of the following periods or visits:

* A 28-day screening period
* Treatment period -

  * Parts A and B: On Day 0, participants will be admitted to hospital for 22-24 hours after injection of ABX-001, which will be administered by a single IV injection as described in the Pharmacy Manual. In the absence of clinical signs and symptoms, participants will be discharged from hospital.
  * Part B: Beginning at Week 3, participants in Part B will receive treatment with pembrolizumab every 3 weeks.

ELIGIBILITY:
Inclusion Criteria-

Participants must satisfy all of the following criteria at the screening visit unless otherwise stated:

1. Participant must be capable of giving consent and at least 18 years of age at the time of signing the informed consent.
2. Participants with advanced/recurrent solid tumors.

   Part A: Participants who have progressed despite standard therapy OR are intolerant of standard therapy, OR for whom no standard therapy exists.

   Part B: Participant has histologically confirmed locally advanced or metastatic disease, who have progressed despite standard therapy OR are intolerant of standard therapy, OR for whom no standard therapy exists. Participant must have received pembrolizumab as approved standard of care and have primary refractory or acquired secondary resistance. Participants must have a tumor lesion amenable to biopsy and must have another lesion that can be followed for response.

   As defined by the Society for Immunotherapy of Cancer:

   Primary resistance/refractory to anti-programmed cell death ligand-1 [anti-PD-(L)1]: minimum drug exposure of 8 to 12 weeks or 2 doses of the immunotherapy with lack of benefit, defined as progressive disease (PD) at the time of the first planned assessment of stable disease (SD) lasting less than 6 months.

   Secondary resistance: participants who experience disease progression following complete response (CR)/partial response (PR) or SD ≥6 months or immunotherapy treatment exposure.
3. Histological or cytological documentation of an advanced solid tumor.
4. Participants are willing to undergo tumor biopsy procedures. For tumor biopsies at screening, it is acceptable if a participant has a biopsy within 3 months from screening and/or during or after the most recent line of therapy (with no intervening anticancer therapy), if there is enough material to fulfil the requirements.
5. Measurable disease per RECIST version 1.1. Palpable lesions that are measurable by radiologic or photographic evaluations may be utilized as the only measurable lesion.
6. Eastern Cooperative Oncology Group performance status 0-1.
7. Life expectancy of at least 12 weeks.
8. Adequate organ functions:

   1. absolute neutrophil count ≥1.5 × 10^9/Liter,
   2. hemoglobin ≥90 g/L,
   3. platelets ≥100 × 10^9/Liter,
   4. lymphocyte count ≥0.5 × 10^9/L (500 / mL)
   5. prothrombin time/international normalized ratio and partial thromboplastin time (unless participant is receiving anticoagulant) <1.5 times Upper limit of normal (ULN),
   6. total bilirubin ≤1.5 times ULN, except for participants with Gilbert's syndrome who must have a total bilirubin <3.0 mg/dL,
   7. aspartate transaminase/ alanine aminotransferase ≤2.5 times ULN, for participants with liver metastases/tumor infiltration ≤5 times ULN,
   8. renal system: creatinine clearance ≥45 mL/min (measured or calculated by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula). Estimated glomerular filtration rate by CKD-EPI >60 mL/min,
   9. endocrine system: thyroid stimulating hormone within normal limits,
   10. cardiac system: ejection fraction ≥50% by echocardiogram.
9. Male or female contraceptive requirements:

   a. Female participants are eligible to participate if they are not either pregnant or breastfeeding, and at least one of the following conditions applies: i. Is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, during the study period (participants receiving monotherapy) or 180 days (participants receiving pembrolizumab) after the last dose of study treatment and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relation to the first dose of study treatment.

   ii. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum, as required by local regulations) within 72 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

   The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

   b. Male participants will agree to use contraception.
10. Participants must be willing and able to communicate and participate in the entire study.
11. Participants must be able and willing to comply with study assessments and study requirements.
12. Participants must be able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions.

Exclusion Criteria -

Participants will be excluded from the study if they satisfy any of the following criteria at the screening visit unless otherwise stated:

1. Malignancy other than disease under study with the exception of those from which the participant has been disease-free for more than 2 years and not expected to affect the safety of the participant or the endpoints of the study. Curatively treated non-melanoma skin cancer is permitted.
2. Symptomatic central nervous system (CNS) metastases or asymptomatic CNS metastases that have required steroids within 2 weeks prior to first dose of study treatment.
3. Participants with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability. Note: Participants with controlled brain metastases will be allowed but must have completed radiotherapy or surgery for CNS metastases >2 weeks prior to study entry. Participants must be neurologically stable, having no new neurologic deficits on clinical examination, and without evidence of progression for at least 4 weeks by repeat imaging (which should be performed during study screening).
4. Active autoimmune disease that has required systemic disease modifying or immunosuppressive treatment within the last 2 years. Replacement therapy (eg, thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
5. Concurrent medical condition requiring the use of systemic immunosuppressive treatment within 28 days before the first dose of study treatment. Physiologic doses of corticosteroids for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids may be continued if the participant is on a stable dose, such as:

   1. Intranasal, inhaled, topical steroids, or local steroid injection (eg, intra-articular injection)
   2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
   3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
6. Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria.
7. History of vasculitis at any time prior to study treatment.
8. Evidence or history of significant active bleeding or severe coagulation dysfunction within the last 6 months prior to receiving the first dose of study treatment.
9. Known human immunodeficiency virus infection, and active and chronic hepatitis B, or hepatitis C.
10. Participants with any kind of active infection, regardless of ongoing systemic treatment.
11. QT interval corrected for heart rate using Fridericia's method >450 msec or QTcF >480 msec for participants with bundle branch block. A QTcF is the QT interval corrected for heart rate according to Fridericia's formula, machine-read or manually over-read.
12. Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
13. Recent history of allergen desensitization therapy within 4 weeks of starting study treatment.
14. History or evidence of cardiovascular risk including any of the following: Recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities including second degree (Type II) or third degree atrioventricular block; cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrolment; clinically uncontrolled hypertension, congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system.
15. Recent (within the past 6 months) history of symptomatic pericarditis.
16. History of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia, or evidence of active, non-infectious pneumonitis. Note: Post-radiation changes in the lung related to prior radiotherapy and/or asymptomatic radiation-induced pneumonitis not requiring treatment may be permitted if agreed by the investigator and sponsor.
17. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
18. Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
19. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other condition that could interfere with the participant's safety, obtaining informed consent, or compliance to the study procedures.
20. Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved with this study, unless prospective institutional review board (IRB)/ethics committee (EC) approval (by chair or designee) is given allowing exception to this criterion for a specific participant.
21. Prior treatment with the following agents:

    1. Checkpoint inhibitors, including Programmed cell death protein - 1 (PD-1), Programmed cell death ligand - 1 (PD-L1), and cytotoxic T-lymphocyte-associated antigen 4 inhibitors within 28 days
    2. Anticancer therapy or investigational therapy within 28 days or 5 half-lives of the drug, whichever is shorter
    3. Prior radiation therapy: permissible if at least 1 non-irradiated measurable lesion is available for assessment according to RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A washout of at least 28 days before start of study treatment for radiation of any intended use to the extremities for bone metastases and 28 days for radiation to the chest, brain or visceral organs is required. Palliative radiation is permissible at any time before or during the study.
22. Receipt of any live vaccine within 30 days of the start of study treatment.
23. Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
24. Toxicity from previous treatment including: Toxicity ≥ Grade 3 related to prior immunotherapy and that led to study treatment discontinuation; toxicity related to prior treatment that has not resolved to ≤ Grade 1 (except alopecia, hearing loss, or ≤ Grade 2 neuropathy or endocrinopathy managed with replacement therapy).
25. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], Granulocyte macrophage colony stimulating factor [GM-CSF], and recombinant erythropoietin) within 14 days before the first dose of study treatment.
26. Major surgery ≤28 days before the first dose of study treatment. Participants must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
27. Known drug or alcohol abuse.
28. Hypersensitivity to the active substance or to any of the excipients of the IMP or checkpoint inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) in the DLT evaluation period | 3 weeks from start of treatment
Incidence and severity of Adverse Events (AEs) throughout the study | Part A: Up to 12 weeks, Part B: Up to 2 years

SECONDARY OUTCOMES:
Objective Responses (OR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and immune RECIST | From start of treatment until progression, death, or end of study, whichever occurs first (Part A: Up to 12 weeks, Part B: Up to 2 years)
Best percentage change from baseline in size of target lesions | From start of treatment until progression, death, or end of study, whichever occurs first (Part A: Up to 12 weeks, Part B: Up to 2 years)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Charite-Universitaetsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Universitaetsklinikum Tuebingen, Tübingen
- Spain (3):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - The START Center for Cancer Care - CIOCC, Madrid